CLINICAL TRIAL: NCT03022045
Title: A Phase 3, Randomized, Open-Label Study to Assess Efficacy and Safety of Two Different Dose Regimens of Risankizumab Administered Subcutaneously in Japanese Subjects With Generalized Pustular Psoriasis or Erythrodermic Psoriasis
Brief Title: A Study to Assess Efficacy and Safety of Two Different Dose Regimens of Risankizumab Administered Subcutaneously in Japanese Subjects With Generalized Pustular Psoriasis or Erythrodermic Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M15-988
Record Dates: First submitted 2017-01-13; First posted 2017-01-16 (Estimated); Results first posted 2019-02-06 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Psoriasis
Keywords: Generalized Pustular Psoriasis; Erythrodermic Psoriasis; risankizumab; Japanese
MeSH Terms: conditions — Psoriasis | interventions — risankizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Risankizumab 75 mg (Experimental): Participants randomized to receive risankizumab 75 mg at Week 0, Week 4, and every 12 weeks up to Week 172.
  Interventions: Drug: risankizumab
- Risankizumab 150 mg (Experimental): Participants randomized to receive risankizumab 150 mg at Week 0, Week 4, and every 12 weeks up to Week 172.
  Interventions: Drug: risankizumab

INTERVENTIONS:
Drug: risankizumab — risankizumab administered by subcutaneous injection
  Other Names: ABBV-066 BI 655066

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of two different dose regimens of risankizumab for Japanese subjects with generalized pustular psoriasis (GPP) or erythrodermic psoriasis (EP).

DETAILED DESCRIPTION:
Safety and efficacy data through 14 December 2017 are included in the interim analysis, which was conducted after all participants completed the Week 28 visit or discontinued from the study.

ELIGIBILITY:
Inclusion Criteria:

For GPP

* Have a diagnosis of GPP for at least 60 days prior to informed consent based on the diagnostic criteria of the Japanese Dermatological Association (JDA). Subjects not fulfilling one of the diagnostic criteria i.e., "accompanying systemic symptoms including fever or malaise" at the time of screening can be entered.
* Subjects with an erythema area with pustules accounting for ≥ 10% of the body surface area (BSA), and with a severity assessment criteria score (JDA total score) specified by the JDA of less than 14.
* Must be candidates for systemic therapy or phototherapy for GPP, as assessed by the investigator.

For EP

* Have a diagnosis of EP prior to informed consent.
* Subjects with an inflammatory erythema area accounting for ≥ 80% of the BSA at screening and at the time of the first administration of the study drug.
* Must be candidates for systemic therapy or phototherapy for EP, as assessed by the investigator.

Exclusion Criteria:

* Previous exposure to risankizumab.
* Currently enrolled in another investigational study or less than 30 days (from screening) since completing another investigational study (participation in observational studies is permitted).

For GPP

* Subjects with active ongoing inflammatory diseases other than GPP that might confound trial evaluations according to investigator's judgment.

For EP

* Subjects with active ongoing inflammatory diseases other than EP that might confound trial evaluations according to investigator's judgment.
* Subject diagnosed with medication-induced or medication-exacerbated EP.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2017-09-17 (Actual); Study Completion 2020-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (9):
- Japan (9):
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Juntendo Univ Urayasu Hosp, Urayasu Shi, Chiba
  - Takagi Dermatological Clinic, Obihiro, Hokkaido
  - Mie University Hospital, Tsu, Mie-ken
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Shizuoka General Hospital, Shizuoka, Shizuoka
  - Tokyo Medical University Hosp, Shinjuku-ku, Tokyo
  - Fukuoka University Hospital, Fukuoka
  - The University of Tokyo Hosp, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Suleiman AA, Khatri A, Oberoi RK, Othman AA. Exposure-Response Relationships for the Efficacy and Safety of Risankizumab in Japanese Subjects with Psoriasis. Clin Pharmacokinet. 2020 May;59(5):575-589. doi: 10.1007/s40262-019-00829-2. PMID 31667790
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/us/clinical-trials/risankizumab_M15-988.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 18 subjects were enrolled; 1 subject failed screening and are excluded from the analyses.
Period: Overall Study
Arm/Group | Risankizumab 75 mg | Risankizumab 150 mg
Started | 9 | 8
Completed (As of the interim analysis data cutoff (14 December 2018)) | 8 | 6
Not Completed | 1 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Risankizumab 75 mg | Risankizumab 150 mg | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (20.76) | 44.1 (20.13) | 48.40 (20.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 8 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Generalized Pustular Psoriasis (GPP) Achieving GPP Clinical Response at Week 16
Description: GPP Clinical Response defined as at least "Slightly Improved" in the overall improvement rating from baseline according to Japanese Dermatological Association (JDA) total score for GPP. The JDA consists of an assessment of skin symptoms (area of skin with erythema, pustules, and edema) on a scale of 0 (none) to 9 (severe) and a systemic symptoms/assessment of test findings (fever, white blood count [WBC], serum C-reactive protein [CRP], and serum albumin) on a scale of 0 (none) to 8 (severe). The JDA total score is the sum of the 2 assessments ranging from 0 (mild) to 17 (severe). The overall improvement rating ranges from Markedly improved (decreased by ≥ 3 points) to Worsened (increased by ≥ 1 point); Slightly improved represents no change in points and ≥ 20% and < 30% reduction of erythema area with pustules compared to baseline, or clinically meaningful improvement in ≥1 other parameters of the severity assessment criteria. Nonresponder imputation (NRI) was used for missing data.
Time Frame: Week 16
Measure: Number; unit: percentage of participants
Groups:
- GPP Risankizumab 75 mg: Participants with generalized pustular psoriasis (GPP) randomized to receive risankizumab 75 mg at Week 0, Week 4, and every 12 weeks up to Week 172.
- GPP Risankizumab 150 mg: Participants with generalized pustular psoriasis (GPP) randomized to receive risankizumab 150 mg at Week 0, Week 4, and every 12 weeks up to Week 172.
Arm/Group | GPP Risankizumab 75 mg | GPP Risankizumab 150 mg
Number analyzed (Participants) | 4 | 4
percentage of participants | 100 | 100

2. Primary Outcome: Percentage of Participants With Erythrodermic Psoriasis (EP) Achieving EP Clinical Response at Week 16
Description: EP Clinical Response, defined as at least "Minimally Improved" in Clinical Global Impression-Global Improvement (CGI-GI) for EP. The CGI-GI is a global assessment by the Investigator of the change in clinical status since the start of treatment. The CGI-GI ratings are as follows: 0 (not assessed), 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse), 7 (very much worse). NRI was used for missing data.
Time Frame: Week 16
Measure: Number; unit: percentage of participants
Groups:
- EP Risankizumab 75 mg: Participants with erythrodermic psoriasis (EP) randomized to receive risankizumab 75 mg at Week 0, Week 4, and every 12 weeks up to Week 172.
- EP Risankizumab 150 mg: Participants with erythrodermic psoriasis (EP) randomized to receive risankizumab 150 mg at Week 0, Week 4, and every 12 weeks up to Week 172.
Arm/Group | EP Risankizumab 75 mg | EP Risankizumab 150 mg
Number analyzed (Participants) | 5 | 4
percentage of participants | 100 | 100

3. Secondary Outcome: Percentage of Participants With GPP Achieving GPP Clinical Response at Week 52
Description: GPP Clinical Response defined as at least "Slightly Improved" in the overall improvement rating from baseline according to JDA total score for GPP. The JDA consists of an assessment of skin symptoms (area of skin with erythema, pustules, and edema) on a scale of 0 (none) to 9 (severe) and a systemic symptoms/assessment of test findings (fever, WBC, serum CRP, and serum albumin) on a scale of 0 (none) to 8 (severe). The JDA total score is the sum of the 2 assessments ranging from 0 (mild) to 17 (severe). The overall improvement rating ranges from Markedly improved (decreased by ≥ 3 points) to Worsened (increased by ≥ 1 point); Slightly improved represents no change in points and ≥ 20% and < 30% reduction of erythema area with pustules compared to baseline, or clinically meaningful improvement in ≥1 other parameters of the severity assessment criteria.
Time Frame: Week 52
Reporting Status: Not Posted, anticipated posting 2022-01

4. Secondary Outcome: Percentage of Participants With EP Achieving EP Clinical Response at Week 52
Description: EP Clinical Response, defined as at least "Minimally Improved" in CGI-GI for EP. The CGI-GI is a global assessment by the Investigator of the change in clinical status since the start of treatment. The CGI-GI ratings are as follows: 0 (not assessed), 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse), 7 (very much worse).
Time Frame: Week 52
Reporting Status: Not Posted, anticipated posting 2022-01

5. Secondary Outcome: Percentage of Participants With GPP Achieving 90% Improvement in Psoriasis Area and Severity Index (PASI) Score (PASI90) at Week 16
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI90 is defined as at least a 90% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100.
Time Frame: Week 16
Measure: Number; unit: percentage of participants
Arm/Group | GPP Risankizumab 75 mg | GPP Risankizumab 150 mg
Number analyzed (Participants) | 4 | 4
percentage of participants | 100 | 75

6. Secondary Outcome: Percentage of Participants With EP Achieving PASI90 at Week 16
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI90 is defined as at least a 90% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100. NRI was used for missing data.
Time Frame: Week 16
Measure: Number; unit: percentage of participants
Arm/Group | EP Risankizumab 75 mg | EP Risankizumab 150 mg
Number analyzed (Participants) | 5 | 4
percentage of participants | 60 | 100

7. Secondary Outcome: Percentage of Participants With GPP Achieving PASI90 at Week 52
Description: as for outcome 5
Time Frame: Week 52
Reporting Status: Not Posted, anticipated posting 2022-01

8. Secondary Outcome: Percentage of Participants With EP Achieving PASI90 at Week 52
Description: as for outcome 5
Time Frame: Week 52
Reporting Status: Not Posted, anticipated posting 2022-01

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 105 days after the last dose of study drug (up to 187 weeks).
Description: TEAEs and SAEs are defined as any AE or SAE with onset or worsening from the time that the first dose of risankizumab is administered until 105 days after the last dose of study drug.
Arm/Group | GPP Risankizumab 75 mg | GPP Risankizumab 150 mg | EP Risankizumab 75 mg | EP Risankizumab 150 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 2/4 | 1/5 | 1/4
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 3/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GPP Risankizumab 75 mg (N=4) | GPP Risankizumab 150 mg (N=4) | EP Risankizumab 75 mg (N=5) | EP Risankizumab 150 mg (N=4)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alcoholic liver disease (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GPP Risankizumab 75 mg (N=4) | GPP Risankizumab 150 mg (N=4) | EP Risankizumab 75 mg (N=5) | EP Risankizumab 150 mg (N=4)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 3 (4) | 3 (4)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2017-01-23): https://cdn.clinicaltrials.gov/large-docs/45/NCT03022045/Prot_001.pdf
  • Statistical Analysis Plan (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/45/NCT03022045/SAP_000.pdf